CLINICAL TRIAL: NCT05993728
Title: Effectiveness of the Body Project to Prevent Eating Disorders in Young Females at Risk: a Randomized Controlled Trial
Brief Title: Virtual Body Project Groups Led by Peers Versus Clinicians
Acronym: v-BP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Karolinska Institutet (Other); Stanford University (Other); Oslo New University College, Norway (Unknown)
Responsible Party: Principal Investigator, Line Wisting, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 609734
Record Dates: First submitted 2023-07-31; First posted 2023-08-15 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Eating Disorders; Body Image
Keywords: Prevention; Body acceptance
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The assessor completing the diagnostic interview will be blinded to the condition the participant is in (at all assessments)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinician-led Body Project (Experimental): Participants randomized to this condition will take part in virtual Body Project groups led by clinicians.
  Interventions: Behavioral: Body Project
- Peer-led Body Project (Experimental): Participants randomized to this condition will take part in virtual Body Project groups led by peers.
  Interventions: Behavioral: Body Project
- Educational control (Active Comparator): Participants randomized to the educational control group will receive educational videos on body image and eating disorders
  Interventions: Behavioral: Psychoeducational control

INTERVENTIONS:
Behavioral: Body Project — The Body Project prevention program is a body acceptance program to promote a healthy body image and prevent eating disorder onset.
  Arms: Clinician-led Body Project; Peer-led Body Project
Behavioral: Psychoeducational control — Participants randomized to the educational control condition will receive videos addressing body image and eating disorders
  Arms: Educational control

SUMMARY:
Eating disorders (EDs) are a group of illnesses associated with significant psychological and physiological consequences. Overall, only 20% of individuals with EDs receive treatment and treatment is effective for only about 25-35% for those who receive care. The development and implementation of effective prevention approaches for those at risk is therefore pivotal. The Body Project is the most effective ED prevention program for at-risk females according to meta-analyses, but reach has been limited since delivery has traditionally been in-person. Further research is warranted to examine cost-effective and easily accessible approaches to increase scalability and potential for broad implementation. With this application, the investigators therefore propose to examine the effectiveness of the Body Project in young females, a high-risk group, with the following main novel aspects: i) virtually-delivered Body Project groups to maximize reach; ii) peer-led versus clinician-led virtually-delivered Body Project groups; iii) the inclusion of objective measures to assess engagement of intervention targets (i.e., mediator).

ELIGIBILITY:
Inclusion Criteria:

* Age 16-25
* Female identifying
* Self-reported body image concerns

Exclusion Criteria:

* Ongoing eating disorder diagnosis requiring treatment or hospitalization

Ages: 16 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Female-identifying
Enrollment: 441 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change over time in eating disorder symptoms | Baseline/pretest, posttest right after intervention (an average of 8 weeks), and at follow-up after 6-months, 1-year, and 2-years
  Assessed with the 28-item self-report Eating Disorder Examination Questionnaire (EDE-Q). Responses range from 0-6, whith higher scores indicating more severe eating disorder psychopathology
Rate of eating disorder onset | Baseline/pretest, 1-year, and at 2-years
  Assessed with the eating disorder diagnostic interview Eating Disorder Assessment-5 (EDA-5). This is a semi-structured clinician-led diagnostic interview, based on the diagnostic criteria in the diagnostic manual DSM-5, and is efficient to determine eating disorder diagnostic status. This outcome will be used to determine proportion of participants with an eating disorder diagnosis.
Change over time in Body dissatisfaction | Baseline/pretest, posttest right after intervention (an average of 8 weeks), and at follow-up after 6-months, 1-year, and 2-years
  Assessed with the 10-item Body Dissatisfaction Scale (BDI; Berscheid et al., 2973) which assesses dissatisfaction with various body parts. Each item is scored on a scale of 1 = extremely dissatisfied to 5 = extremely satisfied. Lower scores indicate greater body dissatisfaction
Change over time in thin-ideal internalization | Baseline/pretest, posttest right after intervention (an average of 8 weeks), and at follow-up after 6-months, 1-year, and 2-years
  Assessed with the 8-item Ideal-Body Stereotype Scale-Revised (Stice et al., 2017) which measures pursuit of the thin ideal. Each item is scored on a scale of 1 = strongly disagree to 5 = strongly agree. Higher scores indicate greater belief in the thin-deal.
Negative affect | Baseline/pretest, posttest right after intervention (an average of 8 weeks), and at follow-up after 6-months, 1-year, and 2-years
  20 negative items from the Positive and Negative Affect Schedule - Revised (PANAS-X) (Watson & Clark, 1992) to measure negative affect. Higher scores indicate higher levels of negative affect. Responses range from 1-5

SECONDARY OUTCOMES:
Change over time in appearance ideals and perceived pressures | Baseline/pretest, posttest right after intervention (an average of 8 weeks), and at follow-up after 6-months, 1-year, and 2-years
  Assessed with the Attitudes Towards Appearance Questionnaire (SATAQ-4R) (Schaefer et al., 2017). A total of 31 items are included, and responses range from 1-5. Higher scores indicate higher levels of internalization/pressures

CONTACTS AND LOCATIONS:
Overall Officials: Line Wisting, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wisting L, Stice E, Ghaderi A, Dahlgren CL. Effectiveness of virtually delivered Body Project groups to prevent eating disorders in young women at risk: a protocol for a randomized controlled trial. J Eat Disord. 2023 Nov 24;11(1):209. doi: 10.1186/s40337-023-00932-7. PMID 38001544